CLINICAL TRIAL: NCT07205640
Title: Effect of Low-Level Laser Therapy Versus Hyaluronic Acid on Wound Healing After First Permanent Molar Extraction in Children.
Brief Title: Improving Healing in Children After Tooth Extraction Using Laser Therapy or Hyaluronic Acid
Acronym: LLLT vs HA
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mona Ali Abd Elhafiz Ali, Bachelor Degree in Oral and Dental Medicine, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: LLLTvsHA-2025
Record Dates: First submitted 2025-08-08; First posted 2025-10-03 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-09

CONDITIONS: Mesh; Healthy Volunteer; Low Level Laser Therapy; Hyaluronic Acid Gel for Preservation the Extraction Socket; Extraction Socket Healing; Badly Decayed Molars; Tooth Extraction Site Healing
Keywords: hyaluronic acid; low level laser therapy; tooth extraction
MeSH Terms: interventions — Low-Level Light Therapy; Hyaluronic Acid

STUDY DESIGN:
Who Masked: Participant
Masking Description: outcome assessors and statistician
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Low-Level Laser Therapy (LLLT) (Experimental): Participants in this arm will receive low-level laser therapy (LLLT) immediately after extraction of the first permanent molar.
  Interventions: Device: Low-Level Laser Therapy
- Hyaluronic Acid (HA) (Experimental): Participants in this arm will receive hyaluronic acid (HA) immediately after extraction of the first permanent molar.
  Interventions: Drug: Hyaluronic Acid (HA)

INTERVENTIONS:
Device: Low-Level Laser Therapy — A 980 nm diode laser will be applied immediately after extraction of the first permanent molar. The laser will be used in continuous mode at 0.5 W, with a total energy of 300 J, applied for 60 seconds at three points around the extraction socket.
  Arms: Low-Level Laser Therapy (LLLT)
Drug: Hyaluronic Acid (HA) — Hyaluronic acid gel will be applied directly into the extraction socket immediately after tooth removal.
  Arms: Hyaluronic Acid (HA)

SUMMARY:
Tooth extraction may be an unpleasant and painful experience for children, Post-extraction wound healing. Low-level laser therapy (LLLT) is a widely used adjuvant treatment for wound healing, resulting in both an increase in cell number and an increase in cell metabolism. HA it is an important component of the extracellular matrix and a constituent of the neural, connective, and epithelial tissues.

DETAILED DESCRIPTION:
Tooth extraction may be an unpleasant and painful experience for children. Pain felt during dental treatment, especially tooth extraction, is the most common complication. Pain management during and after tooth extraction is part of behavioral guidance, especially in pediatric patients.

Post-extraction wound healing and pain perception are related to hostrelated factors such as the patient's immune system, the use of painkillers and antibiotics, the presence of infection in the region, and the atraumatic nature of the procedure. Low-level laser therapy (LLLT) is a widely used adjuvant treatment for wound healing. It is based on the idea that exposure to a specific wavelength can alter cellular behavior, resulting in both an increase in cell number and an increase in cell metabolism. Aside from not having any negative effects, LLLT is an a thermic, photobiological, and nondestructive therapy approach.

HA it is an important component of the extracellular matrix and a constituent of the neural, connective, and epithelial tissues. Among the many biological effects of HA are its functions in cell differentiation, wound healing, inflammation, embryological development, and viscoelasticity.

ELIGIBILITY:
Inclusion Criteria:

1. Children aged from six to ten years.
2. Children of both genders.
3. Children with badly decayed first permanent molar beyond repair and indicated for extraction.
4. Parents acceptance to participate in the study.

Exclusion Criteria:

1. Medically compromised children.
2. Uncooperative children.
3. Children who will not attend the follow up visits

Ages: 6 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 36 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
wound size | 7 days
  Wound size unit of measure : mm (millimeters) (mesiodistal and buccolingual dimension of each socket).

SECONDARY OUTCOMES:
Tissue Color Changes | Day 0, Day 3, and Day 7 post-extraction.
  Gingival color assessed using the Landry, Turnbull, and Howley Index (normal vs inflamed).
  Unit of Measure: Binary (normal / inflamed)
Bleeding Upon Palpation | Day 0, Day 3, and Day 7 post-extraction.
  Presence or absence of bleeding when palpating the extraction site.
  Unit of Measure: Binary (yes / no)
Pus Presence | Day 0, Day 3, and Day 7 post-extraction.
  Presence or absence of pus at the extraction site.
  Unit of Measure: Binary (yes / no)
Pain Level During Application | Immediately after intervention (Day 0).
  Pain assessed using Wong-Baker Faces Pain Rating Scale (0 = no pain, 10 = worst pain).
  (0 = no pain, 10 = worst pain). Higher scores indicate worse outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Mona Ali Abd Elhafiz, BDS, Principal Investigator — Cairo University
Locations (1):
- Faculty Of Oral & Dental Medicine - Cairo University, Giza, EL Menial, Egypt

IPD SHARING:
Plan to Share IPD: No
This is an academic master's degree study. The individual participant data (IPD) will not be shared outside the study team to ensure patient confidentiality. Only aggregate results will be published.

REFERENCES:
- See also: Background reference on low-level laser therapy and wound healing in dentistry. — https://pubmed.ncbi.nlm.nih.gov/39279207/